CLINICAL TRIAL: NCT07119853
Title: The Effect of Microteaching-Enhanced Advanced Life Support Simulation on Students' Teamwork Skills and Satisfaction: A Quantitative Study
Brief Title: Microteaching and Advanced Life Support Simulation: Effects on Student Satisfaction and Teamwork
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Şehriban Serbest (Other)
Responsible Party: Sponsor-Investigator, Şehriban Serbest, Asst. Prof., Acibadem University
Organization: Acibadem University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ATADEK 2025-07/310
Record Dates: First submitted 2025-07-31; First posted 2025-08-13 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Microteaching
Keywords: Nursing student

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The following interventions were applied to the control group;
  1. Pretest: A 10-question pretest was administered before the theoretical training to assess students' knowledge levels prior to Advanced Life Support training.
  2. Theoretical Training: Following the completion of the pretest, participants received "ERC 2021 Adult Advanced Life Support training" in accordance with the European Resuscitation Council 2021 guidelines in two sessions, one before and one after noon. The training duration was 2 hours.
  3. Simulation Training: Five days after the theoretical training, students received simulation training.
  4. Post-test, student satisfaction and self-confidence evaluation: After the simulation, students took their post-test and filled out data collection forms including the student satisfaction and self-confidence scale and the teamwork scale.
- Microteaching (Experimental): In the experimental group, unlike the control group, simulation training was supported by microteaching.
  Microteaching: Students in the experimental group watched the "Advanced Life Support Team Dynamics Video." The video was uploaded to the university's education management system, and a student monitoring report was generated, ensuring that all students could watch it.
  Interventions: Other: Microteaching

INTERVENTIONS:
Other: Microteaching — Students in the experimental group watched the "Advanced Life Support Team Dynamics Video." The video was uploaded to the university's education management system, and a student monitoring report was generated, ensuring that all students could watch it.
  Arms: Microteaching

SUMMARY:
The aim of this study is to evaluate the impact of a microteaching-supported advanced life support simulation on students' teamwork skills and satisfaction.

ELIGIBILITY:
Being a senior nursing student and willing to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Teamwork level measured by Mayo High Performance Teamwork Scale after simulation training | Immediately after the completion of the simulation training session.
  Teamwork was assessed using the Turkish version of the Mayo High Performance Teamwork Scale (MHP-TS). The scale evaluates 16 aspects of team functioning, with each item rated on a 3-point scale: 0 (never), 1 (inconsistent), and 2 (consistent). Total scores range from 0 to 32, with higher scores indicating better teamwork. The scale was administered immediately after the simulation-based advanced life support training supported by microteaching.
Student satisfaction and self-confidence levels measured by the Student Satisfaction and Self-Confidence in Learning Scale after simulation training | Immediately after the simulation training session
  Student satisfaction and self-confidence were assessed using the Turkish version of the Student Satisfaction and Self-Confidence in Learning Scale (SSSCLS). The scale includes two subscales: Satisfaction (5 items) and Self-confidence (8 items). Each item is rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Higher scores indicate greater satisfaction and confidence. The scale was administered immediately after the simulation-based advanced life support training supported by microteaching.

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem Universty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Because I did not receive consent from the participants on this matter.

REFERENCES:
- [Background] Unver V, Basak T, Watts P, Gaioso V, Moss J, Tastan S, Iyigun E, Tosun N. The reliability and validity of three questionnaires: The Student Satisfaction and Self-Confidence in Learning Scale, Simulation Design Scale, and Educational Practices Questionnaire. Contemp Nurse. 2017 Feb;53(1):60-74. doi: 10.1080/10376178.2017.1282319. Epub 2017 Feb 10. PMID 28084900
- [Background] Malec JF, Torsher LC, Dunn WF, Wiegmann DA, Arnold JJ, Brown DA, Phatak V. The mayo high performance teamwork scale: reliability and validity for evaluating key crew resource management skills. Simul Healthc. 2007 Spring;2(1):4-10. doi: 10.1097/SIH.0b013e31802b68ee. PMID 19088602
- [Background] INACSL Standards Committee, Bowler, F., Klein, M. & Wilford, A. (2021, September). Healthcare Simulation Standards of Best PracticeTM Professional Integrity. Clinical Simulation in Nursing, 58, 45-48. https://doi.org/10.1016/j.ecns.2021.08.014.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT07119853/Prot_SAP_ICF_000.pdf